CLINICAL TRIAL: NCT06597305
Title: Twenty-session Cognitive-behavioral Therapy for Adults With Anorexia Nervosa (CBT-20-AN)
Brief Title: Evaluation of a Twenty-session Cognitive-behavioral Therapy With Anorexia Nervosa (CBT-20-AN) Among Adults (18+)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kendra R. Becker, Ph.D., Eating Disorder Clinical and Research Program (EDCRP) Director of Translational Research/Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P002713
Record Dates: First submitted 2024-04-18; First posted 2024-09-19 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CBT-20-AN (Experimental): The single CBT-20-AN arm of this study is experimental, consisting of 20 weekly sessions and one-month, three-month, and six-month follow-ups.
  Interventions: Behavioral: Twenty Session Cognitive-Behavioral Therapy for Anorexia Nervosa (CBT-20-AN)

INTERVENTIONS:
Behavioral: Twenty Session Cognitive-Behavioral Therapy for Anorexia Nervosa (CBT-20-AN) — Twenty session cognitive behavioral therapy for Anorexia Nervosa (CBT-20-AN) is an treatment for Anorexia Nervosa delivered by a mental health clinician. This treatment (CBT-20-AN) lasts just 20 sessions and has been designed to allow individuals with AN to reap the benefits of CBT for eating disorders (up to 40 sessions) in less time, increasing access to care and shortening time to symptom reduction.

SUMMARY:
The study is a clinical trial assessing the efficacy of a new twenty session cognitive behavioral therapy for adults (18+) with anorexia nervosa (AN). It is expected that participants will gain a significant amount of weight and experience a significant decrease in eating disorder psychopathology and behavior from pre- to post- treatment and that this will be retained after 6-months.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients must meet DSM-5 criteria for anorexia nervosa. This diagnosis can be conferred via the EDE 17.0D.
2. Age > 18
3. Patients must be able to provide informed consent and comply with the study procedures.
4. Patients must be able to complete computer-based self-report questionnaires with adequate accommodation, if necessary.
5. Patients must have a primary care physician, Adolescent Medicine physician, or consulting physician with eating disorder expertise at Massachusetts General Hospital/Massachusetts General Brigham network who can provide ongoing medical monitoring while the patient takes part in the study.

Exclusion Criteria:

Patients will be excluded if they exhibit:

1. BMI < 15 or > 19, obtained via patient medical chart or from study 2023P000469 or 2018P002915.
2. HR <55 or >100, obtained via patient medical chart or from study 2023P000469 or 2018P002915.
3. Systolic BP (SBP and DBP) <80 or >160, obtained via patient medical chart or from study 2023P000469 or 2018P002915.
4. Temperature < 96.5 F, obtained via patient medical chart or from study 2023P000469 or 2018P002915.
5. Not eating food by mouth and/or any tube feeding, per EDE
6. Purging > 4x/week, per EDE.
7. Active suicidality (suicidal ideation with intent or plan) to the point that more intensive treatment (i.e. acute hospitalization) is required
8. Active untreated and unstable bipolar disorder (i.e. stable bipolar disorder under care of a psychiatrist is allowed)
9. Psychosis
10. Intellectual disability
11. Any condition that, after the baseline evaluation, is determined to preclude treatment with CBT.
12. Concurrent psychotherapy. Patients must be willing to take a pause from any ongoing psychotherapy in order to focus on CBT-AN-20, which is in alignment with standard clinical care.
13. Symptoms that are not appropriate for outpatient level of care and therefore require a higher level of care (i.e. BMI <15 or purging more than 4x/week)
14. Homicidal ideation
15. Inability to speak English well enough to engage in CBT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Patient weight | Change from study treatment week one to final session, an average of 25 weeks after week one (measured at weekly study treatment sessions), and to the one, three, and six-month follow-up session, up to 11 months after week one.
  Weight collected at each session.
Generalized Anxiety Disorder (GAD-7) | Change from week one of study treatment to post-treatment following final session, an average of 25 weeks after week one (measured at weeks one, six, and twenty), and to one, three, and six-month follow-up sessions, up to 11 months after week one.
  A 7-item scale that measures symptoms of Generalized Anxiety Disorder (GAD), such as feeling anxious or nervous, having trouble relaxing, irritability, and feelings of dread. Scores range from 0 to 21, with higher scores reflecting higher general anxiety.
Patient Health Questionnaire - 9 (PHQ-9) | Change from week one of study treatment to post-treatment following final session, an average of 25 weeks after week one (measured at weeks one, six, and twenty), and to one, three, and six-month follow-up sessions, up to 11 months after week one.
  A 9-item scale that measures symptoms of depression. Scores range from 0 to 27, with higher scores reflecting higher depression.
Eating Disorder Examination Interview (EDE) | Change from baseline assessed at screen visit to post-treatment following final session, an average of 25 weeks after baseline assessment.
  A semi-structured interview designed to assess current eating disorder psychopathology.
Eating Disorder Examination Questionnaire (EDE-Q6) | Change from week one of study treatment to post-treatment following final session, an average of 25 weeks after week one (measured at weeks one, six, and twenty), and to one, three, and six-month follow-up sessions, up to 11 months after week one.
  A 33-item self-report questionnaire that assesses the presence of eating disorders symptoms in the past 28 days. Eating Disorder examination questionnaire (EDE-Q 6.0) Scores range from 0 to 6, with higher scores reflecting higher eating disorder behaviors and attitudes.
Eating Disorder - 15 Scale (ED-15) | Change from study treatment week one to post-treatment following final session, an average of 25 weeks after week one (measured at weekly study treatment session), and to the one, three, and six-month follow-up session, up to 11 months after week one.
  A 15-item self-report measure that assesses eating disorder symptoms and behaviors, designed to measure session-by-session change for clinical and research purposes. Scores range from 0 to 6, with higher scores reflecting higher disordered eating attitudes and behaviors.
Working Alliance Inventory Short (WAI-SR) | Change from week one of study treatment to post-treatment following final session, an average of 25 weeks after week one (measured at weeks one, six, and twenty), and to the six-month follow-up session, up to 11 months after week one.
  A 12-item self-report measure that assess therapeutic alliance between the patient and therapist. (i.e., how comfortable the patient feels with the therapist, how much they trust the therapist, how much they feel the therapist is working towards their desired treatment goals, etc.). Scores range from 5 to 20, with higher scores reflecting higher therapeutic alliance.
General Self-Efficacy Measure-Short Form | Change from week one of study treatment to post-treatment following final session, an average of 25 weeks after week one (measured at weeks one, six, and twenty), and to the six-month follow-up session, up to 11 months after week one.
  A 6-item, short form assessment of the patient's perception of their own general self-efficacy. Scores range from 10 to 40, with higher scores reflecting higher self-efficacy.
Approach/Avoidance of Weighing Questionnaire (AAWQ) | Change from baseline assessed at screen visit to post-treatment following final session, an average of 25 weeks after baseline assessment.
  A 9-item, self-report questionnaire that assesses approach and avoidance weighing tendencies. Items 1-3 are summed to provide the approach weighing tendency subscale and items 4-6 are summed to provide the avoidance weighing tendency subscale, with scores ranging from 3-18. Higher scores on each subscale indicate a higher degree of that subscale's weighing tendency.
Three Factor Eating Questionnaire (TFEQ) - Restriction subscale | Change from baseline assessed at screen visit to session 20 and post-treatment following final session, an average of 20-25 weeks after baseline assessment.
  An 18-item, self-report questionnaire that assesses the presence and severity of restriction.
Eating Disorder Inventory-3 (EDI-3) - Drive for Thinness and Body Dissatisfaction subscales | Change from baseline assessed at screen visit to session 20 and post-treatment following final session, an average of 20-25 weeks after baseline assessment.
  Subscales from the self-report EDI-3 questionnaire that will be used to assess the presence of both drive for thinness and body dissatisfaction. The drive for thinness subscale is 7 items and body dissatisfaction subscale is 10 items.
Clinical Impairment Assessment Questionnaire (CIA) | Change from week one of study treatment to post-treatment following final session, an average of 25 weeks after week one (measured at weeks one, six, and twenty), and to one, three, and six-month follow-up sessions, up to 11 months after week one.
  A 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features.
Quality of life questions | Change from week six of study treatment to post-treatment following final session, an average of 25 weeks after week one (measured at weeks one, six, and twenty), and to one, three, and six-month follow-up sessions, up to 11 months after week one.
  A set of two qualitative questions, developed by the study team, which assess improvements in quality of life since starting treatment ("How has your life improved since beginning treatment?") and areas still needing improvement ("What areas of your life could still be improved?").

CONTACTS AND LOCATIONS:
Locations (1):
- Eating Disorders Clinical and Research Program, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No